CLINICAL TRIAL: NCT03763916
Title: Comparative Study Between Intraoperative Ureteric Dissection and Preoperative Ureteric Stenting in Women With Abnormally Invasive Placenta
Brief Title: Intraoperative Ureteric Dissection vs Preoperative Ureteric Stenting in Women With Abnormally Invasive Placenta
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 44
Record Dates: First submitted 2018-12-03; First posted 2018-12-04 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Placenta Accreta
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intra operative ureteric dissection (Active Comparator): midline abdominal incision extending supraumbilical, incision of the SC tissue, dissection and splitting of the recti, classic midline incision of the uterus [above the site of placental insertion], delivery of the fetus , avoid traction of the placenta, quick closure of the uterus [in presence of the placenta] in one layer, clamping and cutting the round ligament, clamping and cutting the ovarian ligament with ovarian preservation, careful dissection and clamping of the broad ligament varicosities, careful dissection of the post leaflet of the broad ligament until ureter is reached, careful dissection and exposure of both ureter and proper identification of the iliac vessels
  Interventions: Procedure: Ureteric dissection; Procedure: Cesarean hysterectomy
- Preoperative ureteric stenting (Active Comparator): preoperative insertion of ureteric catheters is performed by the urologist in our team just before the start of cesarean hysterectomy. Patient is positioned in lithotomy, cystoscopy [Karl storz] is done to identify the ureteric orifices. ureteric catheters [Roche] are inserted followed by the insertion of Foley's urethral catheter.
  Interventions: Procedure: Preoperative ureteric stenting; Procedure: Cesarean hysterectomy

INTERVENTIONS:
Procedure: Ureteric dissection — clamping and cutting the round ligament, clamping and cutting the ovarian ligament with ovarian preservation, careful dissection and clamping of the broad ligament varicosities, careful dissection of the post leaflet of the broad ligament until ureter is reached, careful dissection and exposure of both ureter and proper identification of the iliac vessels
  Arms: Intra operative ureteric dissection
Procedure: Preoperative ureteric stenting — preoperative insertion of ureteric catheters is performed by the urologist in our team just before the start of cesarean hysterectomy. Patient is positioned in lithotomy, cystoscopy [Karl storz] is done to identify the ureteric orifices. ureteric catheters [Roche] are inserted followed by the insertion of Foley's urethral catheter
  Arms: Preoperative ureteric stenting
Procedure: Cesarean hysterectomy — lateral dissection of the uterus is completed from the pelvic side wall, followed by very CAREFUL BLADDER DISSECTION. Finally clamping of the uterine vessels is done below the level of the placenta with or without complete removal of the cervix. Closure of the uterine stump is performed followed by CAREFUL HEMOSTASIS then closure of the abdomen is performed after leaving two wide bore drains

SUMMARY:
80 Egyptian pregnant female patients will be enrolled in our prospective study. All candidates will have the diagnosis of placenta percreta [confirmed by 2D and 3D ultrasound and Doppler by senior sonographer]. All candidates will be scheduled for cesarean hysterectomy; patients will be randomized into two groups, first group will include 40 patients who will undergo cesarean hysterectomy with intraoperative ureteric dissection, and the second group will include the other 40 patients who will undergo cesarean hysterectomy with preoperative ureteric stenting.

DETAILED DESCRIPTION:
80 pregnant females with the diagnosis of Abnormally invasive placenta [AIP] will be involved in our study [ after proper sample size calculation]. The diagnosis Of AIP will be confirmed by 2D and 3D ultrasound as well as power Doppler evaluation [machine]. Sonographic evaluation will be done and confirmed by senior sonographer in our ACCRETA team.

Patients will be randomized into two groups using closed envelopes after taking written consents; group 1 with intraoperative ureteric dissection and group 2 with preoperative ureteric stenting.

In group 1 cesarean hysterectomy is performed with intra operative ureteric dissection; midline abdominal incision extending supraumbilical, incision of the SC tissue, dissection and splitting of the recti, classic midline incision of the uterus [above the site of placental insertion], delivery of the fetus in presence of a well trained neonatology team, avoid traction of the placenta, quick closure of the uterus [in presence of the placenta] in one layer, clamping and cutting the round ligament, clamping and cutting the ovarian ligament with ovarian preservation, careful dissection and clamping of the broad ligament varicosities, careful dissection of the post leaflet of the broad ligament until ureter is reached, careful dissection and exposure of both ureter and proper identification of the iliac vessels so as to facilitate the ligation of anterior division of internal iliac artery if needed and to avoid any major vascular injury, if unfortunately severe bleeding occurs and rapid surgical intervention is needed. Following ureteric dissection is performed lateral dissection of the uterus is completed from the pelvic side wall, followed by very CAREFUL BLADDER DISSECTION. Finally clamping of the uterine vessels is done below the level of the placenta with or without complete removal of the cervix. Closure of the uterine stump is performed followed by CAREFUL HEMOSTASIS then closure of the abdomen is performed after leaving two wide bore drains.

In group2; preoperative insertion of ureteric catheters is performed by the urologist in our team just before the start of cesarean hysterectomy. Patient is positioned in lithotomy, cystoscopy [Karl storz] is done to identify the ureteric orifices. ureteric catheters [Roche] are inserted followed by the insertion of Foley's urethral catheter. Ureteral catheters are fixed to the Foley's catheter. the ureteric catheters are scheduled for removal immediately postoperative. The patient is then placed in the supine position and sterilization of the abdominal wall is performed and cesarean hysterectomy is performed similarly as in the first group but without ureteric dissection.

The two groups will be carefully studied as regards to incidence of ureteric and bladder injuries, amount of blood loss [measured by weighing towels pre and postoperative; the difference represents the intraoperative blood loss] and the intraoperative timing. Statistical comparison between the rate of complications in each groups will be done. Patients' data will be analyzed statistically using SAS program (SAS, 1996).

ELIGIBILITY:
Inclusion Criteria:

* Parity; multiparas
* Advanced gestational age more than 36 weeks
* Repeated cesarean sections
* Placenta previa
* Abnormally invasive placenta diagnosed and confirmed by senior sonographer

Exclusion Criteria:

* Morbidly obese patient [BMI over 35] Severly anaemic; patients[ Hb less than 8gmLdl] Elderly females [age over 40]
* Inability to insert ureteric stent

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
ureteric injuryoccurance of any type of ureteric injuries including partial , complete transection or inclusion in a ligature | during the operation

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided